CLINICAL TRIAL: NCT02622230
Title: A Randomized, Double-Blind, Placebo-Controlled, Single/ Multiple Dose Study to Assess the Safety , Tolerability, Pharmacokinetics of Mianhuahua Flavonoids Tablets After Oral Administration In Healthy Adult Subjects
Brief Title: Tolerability, Safety and Pharmacokinetic Study Of Mianhuahua Flavonoids Tablets in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinjiang Uygur Pharmaceutical Co., Ltd. (Industry)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XinjiangUP-WY-201501
Record Dates: First submitted 2015-11-23; First posted 2015-12-04 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Uygur Medicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mianhuahua Flavonoids Tablets (Experimental): Mianhuahua Flavonoids Tablets, oral administration
  Interventions: Drug: Mianhuahua Flavonoids Tablets
- Placebo (Placebo Comparator): Placebo, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mianhuahua Flavonoids Tablets — Tolerability Study:
  Period I:Single oral administration,dose-escalation of Mianhuahua Flavonoids Tablets(seven dose groups:0.3g-5.4g) Period II:Repeated oral administration of Mianhuahua Flavonoids Tablets (group 1:MTD（maximum tolerated dose）/1.5g, TID, group 2:depending on the adverse drug reaction,1.8g/1.2g, TID)
  Pharmacokinetic Study:
  Period I:Single oral administration,dose-escalation of Mianhuahua Flavonoids Tablets(six dose groups: 0.9g, 1.8g, 2.7g, 3.6g, 4.5g, 5.4g) Period II:Repeated oral administration of Mianhuahua Flavonoids Tablets (group 1:MTD（maximum tolerated dose）/1.5g, TID, group 2:depending on the adverse drug reaction,1.8g/1.2g, TID)
  Arms: Mianhuahua Flavonoids Tablets
Drug: Placebo — Placebo to match with experimental groups
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability, and to evaluate the pharmacokinetic characteristics of Mianhuahua Flavonoids Tablets after oral administration in healthy adult subjects.

DETAILED DESCRIPTION:
1. Dose-escalation study of single oral administration of Mianhuahua Flavonoids Tablets in healthy adults to assess the safety and tolerability.
2. Multiple-dose study of Mianhuahua Flavonoids Tablets in healthy adults to assess the safety and tolerability.
3. Dose-escalation study of single oral administration of Mianhuahua Flavonoids Tablets in healthy adults to evaluate the pharmacokinetic characteristics
4. Multiple-dose study of Mianhuahua Flavonoids Tablets in healthy adults to evaluate the pharmacokinetics characteristics

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 45 years of age, Body Mass Index (BMI) between 19～24 kg/m2, Weight > or = 50kg
* In good health as judged by the investigator
* Agreed to take effective contraceptive measures during the test and within 6 months after the last drug administration
* Signed informed consent form and fully understood the contents, process and possible adverse reactions of the test

Exclusion Criteria:

* Pregnancy and lactation
* History of kinds of food or drug allergy, or suffering from allergic diseases or allergic constitution
* Presence (in screening stage) or history of the acute/chronic organic diseases or clinical manifestations: Including but not limited to blood system, renal disease, liver disease, endocrine system, respiratory system, digestive system, cardiovascular system, nervous system, mental disease, or any disease and physiological conditions interfering with the results of the test
* with a clinically significant abnormality in routine serological detection: including Hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infected
* History of abuse of drugs, or the result of drug abuse test is positive
* Alcohol intake more than 2 units (1 unit is equal to 12 ounces or 360 ml beer, 5 ounces or 150 ml liquor, 1.5 ounces or 45 ml distilled spirits ) per day on average within 3 months before the test, or the result of alcohol test is positive
* Smoking more than 5 cigarettes per day, or using quite amount of nicotine products within 3 months before the test, or unable to stop smoking during the test
* Excessive consumption of xanthine soda drinks, more than four cups or bottles per day
* With major surgical operations and blood or blood component transfusion within 4 weeks before the test
* Severe blood loss or blood donation more than 400ml within 2 months before the test
* Participation in other drug trials within 3 months before the test
* Usage of any drugs within 2 weeks before the test, or within 5 times of drug eliminated half-life or pharmacodynamics half-life; Vaccination within 4 weeks before the test; Acceptance of biological agents within 4 months before the test
* Be otherwise unsuitable for the study, in the opinion of the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of single and repeated oral administration of Mianhuahua Flavonoids Tablets as measured by the frequency of drug-related clinical adverse events in healthy adults. | Period I: single dose,up to 7 Days;Period II: repeated dose,up to 36 Days
  Safety and tolerability will be evaluated through Composite Metrics：adverse events, vital signs, electrocardiograms, physical exams, and clinical laboratory assessments.

SECONDARY OUTCOMES:
Cmax of single oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 24h
Tmax of single oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 24h
area under curve(AUC) of single oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 24h
t1/2 of single oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 24h
Vd of single oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 24h
Cls of single oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 24h
Css_max of repeated oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 29 days
Css_min of repeated oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 29 days
Tss_max of repeated oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 29 days
area under curve of steady state(AUCss) of repeated oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 29 days
Degree of fluctuation（DF） of repeated oral administration of Mianhuahua Flavonoids Tablets in healthy adults. | up to 29 days

CONTACTS AND LOCATIONS:
Overall Officials: QIU Fu rong, Principal Investigator — Shuguang Hospital affiliated with Shanghai University of TCM